CLINICAL TRIAL: NCT02059525
Title: Treponema Pallidum-specific Proteomic Changes in Patients With Incident Syphilis Infection: an Observational Study in Belgium
Brief Title: Treponema Pallidum-specific Proteomic Changes in Patients With Incident Syphilis Infection
Acronym: SeTPAT
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: SeTPAT
Record Dates: First submitted 2014-02-06; First posted 2014-02-11 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Syphilis
Keywords: observational; Belgium
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- syphilis infected: all patients with a new diagnosis of syphilis, receiving treatment at the Institute of Tropical Medicine

SUMMARY:
This study is part of the Search for a Treponema pallidum Antigen Test (SeTPAT) project to study the proteomic, immunological, serological and clinical changes associated with pre- and post-treatment syphilis infection in a way that could ultimately lead to the development of a new ELISA and rapid diagnostic test of T. pallidum antigenaemia.

The general aim of this prospecive observational cohort study is thus to quantify a set of target proteins with the highest diagnostic potential for the diagnosis of initial T. pallidum infection and T. pallidum persistence. A test which could directly detect the presence of T. pallidum antigens could represent a considerable advance over currently used tests in the diagnosis of initial syphilis infection, its response to therapy and in the diagnosis of syphilis reinfections. This prospective observational cohort study of HIV-positive patients with a new diagnosis of syphilis infection will be conducted at the HIV/Sexually Transmitted Infections (STI) Clinic at the Institute of Tropical Medicine, Antwerp.

DETAILED DESCRIPTION:
This cohort study is part of the Search for a Treponema pallidum Antigen Test (SeTPAT) project to study the proteomic, immunological, serological and clinical changes associated with pre- and post-treatment syphilis infection in a way that will ultimately lead to the development of a new ELISA and rapid diagnostic test of T. pallidum antigenaemia. The general aim of this observational cohort study is thus to quantify a set of target proteins with the highest diagnostic potential for the diagnosis of initial T. pallidum infection and T. pallidum persistence. A test which could directly detect the presence of T. pallidum antigens could represent a considerable advance over currently used tests in the diagnosis of initial syphilis infection, its response to therapy and in the diagnosis of syphilis reinfections.

This prospective observational cohort study of HIV-positive patients with a new diagnosis of syphilis infection will be conducted at the HIV/Sexually Transmitted Infections (STI) Clinic at the Institute of Tropical Medicine, Antwerp (ITM). 120 patients with a new diagnosis of syphilis infection who receive treatment for their syphilis at the ITM and give informed consent, will be recruited; based on the current rate of syphilis diagnosis this should take approximately 18 months. Participants will receive a detailed, standardized clinical assessment, fill out a brief behavioural questionnaire and then be treated with therapy for syphilis according to their stage of disease. In addition to the routine tests performed, if and after they consent to participate in this study, they will have their serum analyzed for a number of other immunological markers. A control group will be recruited, consisting of 30 convenience selected patients who are HIV infected but have no evidence of syphilis (Rapid Plasma Reagin, T. pallidum antigenaemia , or clinical evidence that could be suggestive of syphilis infection) are attending the HIV clinic regularly, who were seen in the same month as one of the acute syphilis cases and who consent to take part in the study. The control group will only undergo the investigations planned for the baseline visit.

Noteworthy, it is hoped that the results of the study will also allow to develop and evaluate the utility of a composite diagnostic rule for the diagnosis of syphilis reinfection.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide written consent
* Prepared to follow the study schedule
* EITHER a diagnosis of a new episode of syphilis - initial or repeat syphilis (Patients group), OR no evidence of past or present syphilis, defined as no clinical or serological evidence of syphilis (Control group).

Exclusion Criteria:

* Use of doxycycline, a macrolide antibiotic or a Beta-lactam antibiotic in the preceding 28 days
* Not willing to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a new diagnosis of syphilis infection who receive treatment for their syphilis at the Institute of Tropical Medicine (ITM), and a control group , consisting of patients who are HIV infected but have no evidence of syphilis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-07; Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
T. Pallidum-specific antigens | Baseline
  Presence/absence and concentration of the T. pallidum-specific antigens

SECONDARY OUTCOMES:
T. pallidum persistence | 6 months pre-penicillin retreatment
  T. pallidum-specific antigens
T. pallidum antigens variation | Any point of suspected treatment failure/reinfection till 24 months
  Changes in T. pallidum-specific antigens, Rapid Plasma Reagin (RPR), T. pallidum antigenaemia (TPA) and Syphilis- immunoglobulin M (IgM)

OTHER OUTCOMES:
Accuracy of screening for Chlamydia trachomatis (CT) and Neisseria gonorrhoea (NG) | 6 months
  CT-positives NG-positives

CONTACTS AND LOCATIONS:
Overall Officials: Chris Kenyon, MD, Principal Investigator — Institute of Tropical Medicine, Belgium
Locations (1):
- Institute of Tropical Medicine, Antwerp, Belgium

REFERENCES:
- [Derived] Osbak KK, Tsoumanis A, De Baetselier I, Van Esbroek M, Smet H, Kenyon CR, Crucitti T. Role of IgM testing in the diagnosis and post-treatment follow-up of syphilis: a prospective cohort study. BMJ Open. 2020 Sep 21;10(9):e035838. doi: 10.1136/bmjopen-2019-035838. PMID 32958482
- [Derived] Van Raemdonck GA, Osbak KK, Van Ostade X, Kenyon CR. Needle lost in the haystack: multiple reaction monitoring fails to detect Treponema pallidum candidate protein biomarkers in plasma and urine samples from individuals with syphilis. F1000Res. 2018 Mar 19;7:336. doi: 10.12688/f1000research.13964.2. eCollection 2018. PMID 30519456
- [Derived] Osbak KK, Van Raemdonck GA, Dom M, Cameron CE, Meehan CJ, Deforce D, Ostade XV, Kenyon CR, Dhaenens M. Candidate Treponema pallidum biomarkers uncovered in urine from individuals with syphilis using mass spectrometry. Future Microbiol. 2018 Oct;13(13):1497-1510. doi: 10.2217/fmb-2018-0182. Epub 2018 Oct 12. PMID 30311792
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/28143443
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/29021408